CLINICAL TRIAL: NCT05613179
Title: Brain Effect Mechanism of Lever Positioning Manipulation on LDH Analgesia Based on Multimodal MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Zhou Xingchen, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSLL-KY-2022-049-01
Record Dates: First submitted 2022-10-24; First posted 2022-11-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Disc Herniation; Multimodal Brain Function; Analgesia Mechanism; Lever Positioning Manipulation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group1 (lever positioning manipulation) (Experimental): Patients with lumbar disc herniation treated by lever positioning manipulation
  Interventions: Procedure: Group1 (lever positioning manipulation)
- Group2 (placebo group) (Active Comparator): Patients with lumbar disc herniation treated by sham lever positioning manipulation
  Interventions: Procedure: Group2 (placebo group)
- Group3 (healthy controls) (No Intervention): Healthy control group without any intervention.

INTERVENTIONS:
Procedure: Group1 (lever positioning manipulation) — The specific lever positioning manipulation is as follows: the patient lies prone at the mouth-open position with muscles relaxed, waist exposed, knees and hips bent, and ankle joints crossed. The practitioner uses the right elbow olecranon to point at the lumbar vertebrae, then hold the patient's two ankle joints in both hands to cause the lumbar vertebra to make hyperextension and flexion movements through the arms and pull the patient backward and upwards hard. When pulling upwards to the trigger point, the practitioner pulls wit lever quickly with a technique and then senses a clatter or looseness at the positioning point. When the practitioner pulls with lever manipulation, the patient is asked to exhale and then inhale at the end of the manipulation.
  Arms: Group1 (lever positioning manipulation)
Procedure: Group2 (placebo group) — The specific sham lever positioning manipulation is as follows: the patient lies prone with his mouth open, muscles relaxed, waist exposed, knees bent at the hip and ankles crossed. The practitioner points to the lumbar spine with the right elbow olecranon, and then holds the patient's two ankles in both hands, so that the lumbar spine through the arm for overextension and flexion, and forcefully pulls the patient back and up. When pulling up to the trigger point, maintain this movement for a short period of time, depending on the patient's endurance, about 1-5 minutes. After finishing, ask the patient to rest in prone position.
  Arms: Group2 (placebo group)

SUMMARY:
In order to further investigate the key brain targets and central response mechanism characteristics of analgesia, the dominant disease of LDH was taken as the object of this study, which was divided into operation group, comfort group and healthy subjects group. Firstly, DTI probabilistic tracking method was used to detect the changes of the brain white matter in each group. Then, the low-frequency amplitude (mfalff) and local consistency (ReHo) of each group were compared by fMRI scanning imaging technology, and the features of local brain functional connectivity (FC) of pain matrix related brain regions as seed points were analyzed. Finally, MRS Technique was used to detect the brain signals of related metabolites glutamic acid (Glu) and 1-aminobutyric acid (GABA), so as to elucidate the network regulation of lever-positioning operation on the analgesic brain effect of LDH and the biochemical mechanism of central nervous system. This multimodal MRI technique provides biological basis for the clinical application of lever localization in LDH.

ELIGIBILITY:
Inclusion Criteria:

1. patients suffering from low back pain and/or radicular leg pain;
2. persistent pain for at least six months that was nonresponsive to conservative treatments;
3. at least one epidural or facet joint corticosteroid injection in the last past year without pain relief or with an improvement in pain of less than two months.
4. Lumbar protrusion level discopathy on MRI corresponding to the level of pain.
5. No interventional pain treatment was applied within the last three months and patients needed a pain score equal or greater than four on the visual analogic scale (VAS).

   -

   Exclusion Criteria:

1.patients with motor deficits, systemic infection, coagulation disorders, pregnancy； 2.VAS pain score lower than four； 3.Patients with any other condition that prevents an MRI scan from being performed.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | up to one month
  Pain intensity was evaluated by means of a visual analogue scale (VAS) [10-point visual analogue scale: 0 = no pain; 10 = very severe pain].
Japanese Orthopaedic Association Scores (JOA) | up to one month
  Japanese Orthopaedic Association Scores (JOA), ranging from 0 (worst) to 100 (best), was used to evaluate the clinical state.
Amplitude of Low-Frequency Fluctuation (ALFF) | up to one month
  The ALFF measures the activity of neurons in the brain that are not affected by external factors.
Regional Homogeneity (ReHo) | up to one month
  The ReHo measures the consistency of the local functional activities of the brain's various regions.
Functional Connectivity (FC) | up to one month
  The FC represents the strength Of functional connections between brain regions, and can reflect the temporal correlation between the Region Of Interest (ROI) and the whole brain networking function.
Diffusion Tensor Imaging (DTI) | up to one month
  The DTI is used to look at images of white matter fiber structures in the brain.
Magnetic Resonance Spectrum （MRS） | up to one month
  The MRS Is the only technology capable of non-invasive quantitative detection of brain substance changes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-zhen Lv, Dr., Study Director — The Third Clinical Medical College of Zhejiang Chinese Medical University, Hangzhou, 310053, China
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Zhou XC, Chen LH, Wu S, Wang KZ, Wei ZC, Li T, Huang YS, Hua ZH, Xia Q, Lv ZZ, Lv LJ. Brain effect mechanism of lever positioning manipulation on LDH analgesia based on multimodal MRI: a study protocol. BMC Complement Med Ther. 2024 Jun 24;24(1):246. doi: 10.1186/s12906-024-04549-4. PMID 38915038